CLINICAL TRIAL: NCT01256099
Title: Guided Internet-treatment for Insomnia. Treatment Effects, Health Economics and Interaction With Depression
Brief Title: Internet-CBT for Insomnia
Acronym: IpsyInsomni
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Region Stockholm (Other Government)
Responsible Party: Principal Investigator, Viktor Kaldo, Principal Investigator, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2009/1810-31/3
Record Dates: First submitted 2010-10-12; First posted 2010-12-08 (Estimated); Last update posted 2015-04-03 (Estimated); Status verified 2015-04

CONDITIONS: Insomnia; Depression
Keywords: Self-help treatment; Internet treatment; CBT; Prevention; Comorbidity
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Guided Internet-CBT for insomnia (Experimental)
  Interventions: Behavioral: Therapist guided Internet-CBT for insomnia
- Control treatment (Placebo Comparator)
  Interventions: Behavioral: Brief Internet-CBT for insomnia, without support
- Guided Internet-CBT for insomnia (9) (Experimental): (9 weeks instead of 8)
  Interventions: Behavioral: Therapist guided Internet-CBT for insomnia
- Guided Internet-CBT for depression (Active Comparator)
  Interventions: Behavioral: Therapist Guided Internet-CBT for depression

INTERVENTIONS:
Behavioral: Therapist guided Internet-CBT for insomnia — An 8 week long, structured self-help program with weekly reports to, and feedback from, a CBT therapist over the Internet. Includes traditional CBT-methods for insomnia
  Arms: Guided Internet-CBT for insomnia; Guided Internet-CBT for insomnia (9)
Behavioral: Brief Internet-CBT for insomnia, without support — No support and less text, not including the CBT-methods that are presumed to be most effective to reduce Insomnia symptoms
  Arms: Control treatment
Behavioral: Therapist Guided Internet-CBT for depression — An 9 week long, structured self-help program with weekly reports to, and feedback from, a CBT therapist over the Internet. Includes traditional CBT-methods for depression. Information and methods regarding sleep difficulties removed
  Arms: Guided Internet-CBT for depression

SUMMARY:
This study includes two sub-trials.

In trial 1 patients suffering from insomnia but not meeting the criteria for depression are randomised to either therapist guided Internet-based CBT for insomnia or to a control group with a non-guided, brief self-help program that acts as a placebo control. The primary purpose is to evaluate reduction in Insomnia severity (compared to placebo) after treatment and at follow-ups at 6-month, 1 year and 3 years. Secondary purpose is to evaluate the costeffectiveness of the treatment and to evaluate if the insomnia treatment has a preventive effect on future depressive episodes. Recruitment is done through mass media and includes all regions of Sweden. Initial assessment based on questionnaires and telephone interviews.

Trial 2 includes patients suffering from both Insomnia and depression. Randomization is done between either CBT for insomnia or CBT for depression (both Internet-based) to evaluate each respective treatment's effect on both insomnia and depression. The patients need for further treatment after the initial one will be measured and used as a secondary outcome. Recruitment is done through mass media but only citizens in the Stockholm area are included since the initial assessment are based on both questionnaires and telephone interviews as well as a visit at a psychiatrist located at the Internet psychiatry clinic in Stockholm.

Both trials will include health economic data and analysis. For the longer follow-up periods (1 and 3 years), registers will be used to analyse consumption of sleep medication and antidepressants as well as general health care utilization.

ELIGIBILITY:
Inclusion Criteria:

* Clinical level of Insomnia (more than 10 on ISI)
* Meets criteria for Insomnia according to DSM-IV-TR
* Enough language skills
* Only Trial 2: Meets criteria for Major Depressive Disorder according to DSM-IV-TR

Exclusion Criteria:

* Sleep disorders requiring other treatment
* High consumption of alcohol/drugs that affect sleep
* Started to use or changed the dose of antidepressant drug during the last 2 months
* Somatic or psychiatric conditions requiring acute care
* Working night shifts
* Only Trial 1: Meets criteria for Major Depressive Disorder according to DSM-IV-TR

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 191 (Actual)
Dates: Start 2010-01; Primary Completion 2014-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Insomnia Severity Index (ISI) | Post-treatment (9 weeks)
  7-item, self-rated questionnaire measuring insomnia severity. Bastien, C. H., Vallières, A., & Morin, C. M. (2001). Validation of the Insomnia Severity Index as an outcome measure for insomnia research. Sleep Medicine, 2, 297-307.
MADRS-S | Post-treatment (9 weeks)
  The use of two primary outcomes are motivated since the purpose is to look at effects on both insomnia and depression. In trial 1 the former is used to predict the latter, and in Trial 2 the patientents suffer from both conditions.
  The MADRS-S is a 9-item self-rated measure of depression severity and screens for suicidality.
  Mattila-Evenden, M., Svanborg, P., Gustavsson, P., & Åsberg, M. (1996). Determinants of self-rating and expert rating concordance in psychiatric out-patients, using the affective subscales of CPRS. Acta Psychiatr Scand, 94, 386-396.
ISI | 6-month follow-up
ISI | 1-year follow-up
ISI | 3-years follow-up
MADRS-S | 6-month follow-up
MADRS-S | 1-year follow-up
MADRS-S | 3-years follow-up

SECONDARY OUTCOMES:
Sleep Diary | Same as primary outcomes
  One week of self-ratings on a number of sleep parameters, resluting in measures of sleep latency, total sleep time, sleep efficacy, number of nighttime awakenings, subjecitve sleep quality and daytime functioning
Trimbos and Institute of Medical Technology Assessment Cost Questionnaire for Psychiatry (TIC-P) | Same as Primary outcomes
  Health economic questionnaire evalutation cost for health care, abscence of work capacity and related costs.
  Hakkaart-Van Roijen, L.,Van Straten, A., & Donker, M. (2002). Manual: Trimbos/iMTA Questionnaire for Costs Associated with Psychiatric Illness. Rotterdam: Erasmus University
EQ-5D | Same as primary outcomes
  General quality of life measure to complement the TIC-P in health economic analysis.
  Hinz, A., Klaiberg, A., Brahler, E., & Konig, H.H. (2006). The Quality of Life Questionnaire EQ-5D: modelling and norm values for the general population. Psychother.Psychosom.Med.Psychol., 56, 42-48.

CONTACTS AND LOCATIONS:
Locations (1):
- Karolinska Institutet, Stockholm, Sweden

REFERENCES:
- [Derived] Kraepelien M, Blom K, Forsell E, Hentati Isacsson N, Bjurner P, Morin CM, Jernelov S, Kaldo V. A very brief self-report scale for measuring insomnia severity using two items from the Insomnia Severity Index - development and validation in a clinical population. Sleep Med. 2021 May;81:365-374. doi: 10.1016/j.sleep.2021.03.003. Epub 2021 Mar 16. PMID 33813233
- [Derived] Blom K, Jernelov S, Ruck C, Lindefors N, Kaldo V. Three-Year Follow-Up Comparing Cognitive Behavioral Therapy for Depression to Cognitive Behavioral Therapy for Insomnia, for Patients With Both Diagnoses. Sleep. 2017 Aug 1;40(8). doi: 10.1093/sleep/zsx108. PMID 28655183
- [Derived] Blom K, Jernelov S, Ruck C, Lindefors N, Kaldo V. Three-Year Follow-Up of Insomnia and Hypnotics after Controlled Internet Treatment for Insomnia. Sleep. 2016 Jun 1;39(6):1267-74. doi: 10.5665/sleep.5850. PMID 27091535
- [Derived] Blom K, Jernelov S, Kraepelien M, Bergdahl MO, Jungmarker K, Ankartjarn L, Lindefors N, Kaldo V. Internet treatment addressing either insomnia or depression, for patients with both diagnoses: a randomized trial. Sleep. 2015 Feb 1;38(2):267-77. doi: 10.5665/sleep.4412. PMID 25337948
- See also: The public page of the Internet-CBT treatment platform — http://www.internetpsykiatri.se